CLINICAL TRIAL: NCT00004068
Title: Treatment of Newly Diagnosed High-Grade Gliomas in Patients Ages Greater Than or Equal to 3 and Less Than or Equal to 21 Years With a Phase II Irinotecan Window Followed by Radiation Therapy and Temozolomide
Brief Title: Irinotecan Followed by Radiation Therapy and Temozolomide in Treating Children With Newly Diagnosed Brain Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067271; P30CA021765 (NIH); SJCRH: SJHG98; SPRI-P-00112; NCI-G99-1577
Record Dates: First submitted 1999-12-10; First posted 2003-05-08 (Estimated); Last update posted 2011-10-04 (Estimated); Status verified 2011-10

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood high-grade cerebral astrocytoma; childhood high-grade cerebellar astrocytoma; childhood oligodendroglioma; untreated childhood brain stem glioma; untreated childhood cerebellar astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Oligodendroglioma | interventions — Irinotecan; Temozolomide; Radiotherapy

INTERVENTIONS:
Drug: irinotecan hydrochloride
Drug: temozolomide
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining chemotherapy with radiation therapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of irinotecan followed by radiation therapy and temozolomide in treating children who have newly diagnosed brain tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the efficacy of adjuvant irinotecan in children with newly diagnosed high grade gliomas, brain stem glioma, or high risk grade II astrocytomas in terms of complete and partial response rate in patients with postoperative measurable disease, and in terms of the rate of freedom from recurrence in patients with no postoperative measurable disease.
* Determine the 3 year overall and progression free survival rates in this patient population when treated with adjuvant irinotecan followed by radiotherapy and temozolomide.
* Assess the hematopoietic toxicity of temozolomide following local radiotherapy in this patient population.

OUTLINE: Patients receive postoperative irinotecan IV over 60 minutes daily for 5 days on weeks 1-2. Treatment repeats every 3 weeks for 2 courses. Following completion of irinotecan and if appropriate, patients may undergo a second surgical resection.

Within 2 weeks following completion of chemotherapy or within 4 weeks of following a second resection, patients receive image guided external beam radiotherapy 5 days per week for 6 weeks. Patients with residual tumor less than 3.5 cm in maximal diameter may undergo boost radiosurgery.

At 4 weeks following completion of radiotherapy, patients receive oral temozolomide for 5 days. Treatment repeats every 3 weeks for 6 courses.

Patients are followed every 3 months for 2 years, then every 4 months for 3 years.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed newly diagnosed brain tumors

  * Grade III or IV disease:

    * Glioblastoma multiforme
    * Anaplastic astrocytoma
    * Anaplastic oligodendroglioma
    * Anaplastic pleomorphic xanthoastrocytoma
    * Anaplastic or malignant oligoastrocytoma
    * Gemistocytic astrocytoma
    * Malignant glioma
  * Grade II glial tumors in unfavorable locations (i.e., imaging evidence of gliomatosis cerebri and/or bithalamic involvement)
  * Diffuse pontine gliomas with greater than 2/3 involvement of the pon

PATIENT CHARACTERISTICS:

Age:

* 3 to 21

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 2,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin greater than 8.0 g/dL

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT less than 5 times normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* Prior corticosteroids allowed

Radiotherapy:

* No prior radiotherapy

Surgery:

* No more than 28 days since prior definitive surgery for brain tumor

Other:

* Concurrent anticonvulsants allowed

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 53 (Actual)
Dates: Start 1999-03; Primary Completion 2003-04 (Actual); Study Completion 2003-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amar Gajjar, MD, Study Chair — St. Jude Children's Research Hospital
Locations (1):
- Saint Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- [Result] Broniscer A, Chintagumpala M, Fouladi M, Krasin MJ, Kocak M, Bowers DC, Iacono LC, Merchant TE, Stewart CF, Houghton PJ, Kun LE, Ledet D, Gajjar A. Temozolomide after radiotherapy for newly diagnosed high-grade glioma and unfavorable low-grade glioma in children. J Neurooncol. 2006 Feb;76(3):313-9. doi: 10.1007/s11060-005-7409-5. PMID 16200343
- [Result] Broniscer A, Iacono L, Chintagumpala M, Fouladi M, Wallace D, Bowers DC, Stewart C, Krasin MJ, Gajjar A. Role of temozolomide after radiotherapy for newly diagnosed diffuse brainstem glioma in children: results of a multiinstitutional study (SJHG-98). Cancer. 2005 Jan 1;103(1):133-9. doi: 10.1002/cncr.20741. PMID 15565574
- [Result] Broniscer A, Chintagumpala M, Bowers D, et al.: Upfront protracted irinotecan (CPT-11) followed by radiotherapy (RT) and temozolomide (TMZ) in the treatment of children with newly diagnosed high-grade glioma (HGG) and unfavorable low-grade glioma (LGG): results of a multi-institutional study (SJHG-98). [Abstract] Neuro-Oncology 6 (4): TP-01, 385, 2004.
- See also: St. Jude Children's Research Hospital — http://www.stjude.org